CLINICAL TRIAL: NCT00282074
Title: Prospective Trial to Evaluate Changes in Spermatogram Following Bilateral Laparoscopic Inguinal Hernia Repair in Males in the Fertility Age
Brief Title: Evaluating Changes in Spermatogram Following Bilateral Laparoscopic Inguinal Hernia Repair in Fertile Males
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SHEBA-05-3945-JK-CTIL
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2007-01-24 (Estimated); Status verified 2007-01

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

INTERVENTIONS:
Procedure: laparoscopic bilateral hernia repair

SUMMARY:
In this prospective open armed study we aim to see if bilateral hernia repair using a mesh alters the spermatogram (sperm count) or testicular volume.

ELIGIBILITY:
Inclusion Criteria:

* Males ages 18-40 years, undergoing bilateral laparoscopic hernia repair, who agree to have a sperm test both prior to and following surgery.

Exclusion Criteria:

* History of prostatic surgery, testicular surgery, azospermia on first spermatogram, single testis, patients after chemotherapy, patients receiving hormonal therapy, patients receiving alpha blockers for any indication, patients who are receiving or received oral antifungal therapy six months prior to surgery

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kuriansky, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel